CLINICAL TRIAL: NCT04847427
Title: Recovery Kinetics of Muscle Performance, Muscle Damage and Neuromuscular Fatigue After Different Protocols of Power Training
Brief Title: Recovery Kinetics After Different Power Training Protocols (PTRecovery)
Acronym: PTRecovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Power training - Recovery
Record Dates: First submitted 2021-02-10; First posted 2021-04-19 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Core Exercises Training; Structural Exercises Training; Accentuated Eccentric Exercises Training; Control Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Core exercises training (Experimental): Participants will perform 4 core exercises
  Interventions: Other: Core exercises training
- Structural exercises training (Experimental): Participants will perform 4 structural (Olympic lifting) exercises
  Interventions: Other: Structural exercises training
- Accentuated eccentric exercises training (Experimental): Participants will perform 4 exercises with eccentric loading
  Interventions: Other: Accentuated eccentric exercises training
- Control trial (Experimental): Participants will perform all the measurements that are comprised in the experimental conditions without performing any exercise protocol
  Interventions: Other: Control trial

INTERVENTIONS:
Other: Core exercises training — Participants will perform:
  1. Squats, 4 sets of 5 repetitions at 60% 1RM
  2. Deadlifts, 4 sets of 5 repetitions at 60% 1RM
  3. Lunges, 4 sets of 5 repetitions at 60% 1RM
  4. Step ups, 4 sets of 5 repetitions at 60% 1RM
  Arms: Core exercises training
Other: Structural exercises training — Participants will perform:
  1. Snatch, 4 sets of 5 repetitions at 60% 1RM
  2. Hang clean, 4 sets of 5 repetitions at 60% 1RM
  3. Push jerk, 4 sets of 5 repetitions at 60% 1RM
  4. Split push jerk, 4 sets of 5 repetitions at 60% 1RM
  Arms: Structural exercises training
Other: Accentuated eccentric exercises training — Participants will perform:
  1. Deadlifts - squat jump, 4 sets of 5 repetitions at 30% body mass (BM)
  2. Step down - squat jump, 4 sets of 5 repetitions at 30% BM
  3. Step down - lunges, 4 sets of 5 repetitions at 30% BM
  4. Bulgarian squat jumps, 4 sets of 5 repetitions at 30% BM
  Arms: Accentuated eccentric exercises training
Other: Control trial — Participants will perform all the measurements that are comprised in the experimental conditions without performing any exercise protocol
  Arms: Control trial

SUMMARY:
Muscle power is one of the most important parameters in almost every athletic action, expressing the ability of the human muscle to produce great amounts of force with the greatest possible speed. For enhancing their muscle power, athletes comprise several resistance training programs as part of their training. However, muscle power training comprises of eccentric muscle actions, which, especially when unaccustomed, can lead to exercise-induced muscle damage and deterioration of muscle performance. Nevertheless, despite the fact that muscle power training comprises eccentric muscle actions, and consequently can lead to muscle injury and muscle performance reduction during the following days, the recovery kinetics after acute muscle power training have not been adequately studied. However, information regarding the recovery of the muscles after a power training protocol, is critical for the correct design of a training microcycle, and the reduction of injury risk. The aim of the present study is to investigate the muscle injury provoked after acute muscle power training using three different power training exercise protocols. Additionally, the effect of these protocols on muscle performance and neuromuscular fatigue indices will be examined.

DETAILED DESCRIPTION:
Muscle power is one of the most important parameters in almost every athletic action, and expresses the ability of the human muscle to produce great amounts of force with the greatest possible speed. Thus, muscle power is critical for high performance in athletic actions such as jumping, throwing, change of direction and sprinting. For enhancing their muscle power, athletes comprise several resistance training programs as part of their training. Core exercises as well as Olympic lifting has been used in muscle power training. The loads that are applied regarding the accomplishment of the most favorable power production are varying. Training load of 0% 1RM has been reported to favor power production at the countermovement squat jump, while loads of 56% 1RM and 80% 1RM, favored the power production at squat and clean, respectively. In the recent years, accentuated eccentric training has been proposed as a new training method for the enhancement of muscle power. This method emphasizes in the eccentric component of the muscle contraction, and there is evidence supporting the greater production of muscle force after accentuated eccentric training compared with the typical resistance exercise training method. Taking the above into consideration, muscle power training comprises of eccentric muscle actions, and the magnitude of the eccentric component depends on the emphasis that is given on the concentric or eccentric action, respectively, of the muscles during the exercises. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD). Although concentric and isometric exercise may also lead to muscle injury, the amount of damage after eccentric muscle contractions is greater. EIMD, amongst others, is accompanied by increased levels of creatine kinase (CK) into the circulation, increased delayed onset of muscle soreness (DOMS), reduction of force production, reduction of agility and speed. Despite the fact that muscle power training comprises eccentric muscle actions and consequently can lead to muscle injury and muscle performance reduction during the following days, the recovery kinetics after acute muscle power training protocols have not been adequately studied. However, information regarding the recovery of the muscles after a power training protocol is critical for the correct design of a training microcycle, and the reduction of injury risk.

The aim of the present study is to investigate the muscle injury provoked after acute muscle power training using three different power training exercise protocols. Additionally, the effect of these protocols on muscle performance and neuromuscular fatigue indices will be examined.

According to a preliminary power analysis, a number of 8 - 10 participants is needed for significant differences to be observed at the variables that will be examined (α = 0.90). Thus, 10 participants will be included at the present study.

The study will be performed in a randomized, cross over, repeated measures design. During their 1st - 4th visit, all participants will sign an informed consent (1st visit) after they will be informed about all the benefits and risks of the study and they will fill and sign a medical history form. Participants will be instructed by a dietitian how to record a 7-days diet recall to ensure that they do not consume in greater extent nutrients that may affect EIMD and fatigue (e.g. antioxidants, amino acids, etc.) and to ensure that the energy intake during the trials will be the same. Subsequently, participants will have to be familiarized with the exercises that will be used during the three power training protocols, as well as with the measurements that will be used for the evaluation of performance indices.

During the 5th, 6th, 7th and 8th visit, baseline assessments will be performed. Fasting blood samples will be collected in order to estimate muscle damage concentration markers. Assessment of body mass and body height, body composition, and aerobic capacity (VO2max), will be performed. Squat jump and countermovement jump will be performed on a force platform to assess jump height, ground reaction force, peak and mean power, vertical stiffness and peak rate of force development; at the same time, peak and mean normalized EMG during the concentric phase of the squat jump, and during eccentric and concentric phases of the counter movement jump, for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles will be assessed. The peak concentric, eccentric and isometric isokinetic torque of the knee flexors and knee extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60°/sec. Maximal voluntary isometric contraction (MVIC) of the knee extensors at 65° in both limbs, as well as the fatigue rate during MVIC through the percent drop of peak torque between the first and the last three seconds of a 10-sec MVIC.

During their 9th visit, participants will be randomly assigned into one of the four different conditions of the study design: a) Core exercises protocol, b) Structural exercises protocol, c) Accentuated eccentric load exercises protocol, d) Control Condition. Prior to each experimental protocol, assessment of DOMS in the knee flexors and knee extensors of both limbs, as well as blood lactate assessment will be performed. Field activity will be continuously recorded during the sprint training protocols using global positioning system (GPS) technology. Heart rate will be continuously recorded during the sprint training protocols using heart rate monitors. Additionally, DOMS of knee flexors and knee extensors, peak concentric, eccentric and isometric isokinetic torque, squat and countermovement jump height, as well as ground reaction force, peak and mean power, vertical stiffness and peak rate of force development during squat and countermovement jump, alongside with peak and mean normalized EMG during the concentric phase of the squat jump, and during eccentric and concentric phases of the counter movement jump, for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles will be assessed immediately after, 24h, 48h and 72h after the end of the trial. MVIC of the knee extensors of both limbs, as well as the fatigue rate during MVIC will also be assessed at 1h, 2h and 3h, as well as 24h, 48h, and 72h (10th, 11th and 12th visit) after the end of the trial. Blood lactate will also be assessed at 4 min, while creatine kinase at 24h, 48h, and 72h after the end of the trial. The exact same procedure (13rd - 16th visit, 17th - 20th visit, 22nd - 24th visit) will be repeated for the remaining three conditions. A 7-day wash out period will be mediated between trials.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year experience in strength exercises
* Absense of musculoskeletal injuries (≥ 6 months)
* Abstence from use of ergogenic supplements or other drugs (≥ 1 month)
* Abstence from participation at exercise with eccentric component (≥ 3 days)
* Abstence from alcohol and energy drings consumption before each experimental trial

Exclusion Criteria:

* Less than 1 year experience in strength exercises
* Musculoskeletal injuries (≤ 6 months)
* Use of ergogenic supplements or other drugs (≤ 1 month)
* Participation at exercise with eccentric component (≤ 3 days)
* Alcohol and energy drings consumption before the experimental trials

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in CK in blood | Baseline (pre), 4 minutes post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  Creatine kinase will be measured in plasma using a biochemical analyzer
Change in delayed onset of muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs | Baseline (pre), 4 minutes post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  Participants will perform three repetitions of a full squat movement, and rate their soreness level in knee flexors and extensors on a visual analog scale from 1 to 10 (VAS, with "no pain" at one end and "extremely sore" at the other), using palpation of the belly and the distal region of relaxed knee extensors and flexors.
Change in blood lactate | Baseline (pre), 4 minutes post-trial
  Blood lactate will be measured in capillary blood with a hand-portable analyzer
Change in squat jump height | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Squat jump height will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate, yet time-synchronized measurement of the jump height for each leg
Change in ground reaction force (GRF) during squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  GRFwill be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate, yet time-synchronized measurement of the jump height for each leg
Change in peak power during squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Peak power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate, yet time-synchronized measurement of the jump height for each leg
Change in mean power during squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate, yet time-synchronized measurement of the jump height for each leg
Change in vertical stifness during squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Vertical stifness will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate, yet time-synchronized measurement of the jump height for each leg
Change in peak normalized EMG during the concentric phase of the squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles.
Change in mean normalized EMG during the concentric phase of the squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles.
Change in countermovement jump height | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Countermovement jump height will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in ground reaction force (GRF) during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Ground reaction force will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak power during countermovement jump test | Baseline (pre), post-, 24h post-, 48h post-, 72h post-trial
  Peak power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in mean power during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in vertical stifness during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Vertical stifness will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak rate of force development during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Vertical stifness will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak normalized EMG during the eccentric and concentric phases of the countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles.
Change in mean normalized EMG during the eccentric and concentric phases of the countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles.
Change in concentric peak torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Concentric peak torque will be measured on an isokinetic dynamometer
Change in eccentric peak torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Eccentric peak torque will be measured on an isokinetic dynamometer
Change in isometric peak torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Eccentric peak torque will be measured on an isokinetic dynamometer
Change in maximal voluntary isometric contraction (MVIC) during 10 seconds | Baseline (pre), 1 hour post-, 2 hours post-, 3 hours post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  MVIC will be measured on an isokinetic dynamometer
Change in fatigue rate during maximal voluntary isometric contraction (MVIC) | Baseline (pre), 1 hour post-, 2 hours post-, 3 hours post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  Fatigue rate during MVIC will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-second maximal isometric contaction
Differences in field activity between the three different power training protocols | During each power training protocol
  Field activity will be continuously recorded during the power training protocols using global positioning system (GPS) technology
Change in heart rate between the three different power training protocols | During each power training protocol
  Heart rate will be continuously recorded during during the power training protocols using heart rate monitors

SECONDARY OUTCOMES:
Body weight | Baseline
  Body weight will be measured on a beam balance/stadiometer
Body height | Baseline
  Body height will be measured on a beam balance/stadiometer
Body mass index (BMI) | Baseline
  BMI will be calculated from the ratio of body mass/ body height squared
Maximal oxygen consumption (VO2max) | Baseline
  Maximal oxygen consumption will be measured by open circuit spirometry via breath by breath method
Body fat | Baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry
Lean body mass | Baseline
  Lean body mass will be measured by using Dual-emission X-ray absorptiometry
Dietary intake | Baseline
  Dietary intake will be assessed using 7-day diet recalls

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Principal Investigator — Department of Physical Education and Sport Science, University of Thessaly
Locations (1):
- Chariklia K. Deli, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarkson PM, Byrnes WC, McCormick KM, Turcotte LP, White JS. Muscle soreness and serum creatine kinase activity following isometric, eccentric, and concentric exercise. Int J Sports Med. 1986 Jun;7(3):152-5. doi: 10.1055/s-2008-1025753. PMID 3733311
- [Background] Deli CK, Fatouros IG, Paschalis V, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. A Comparison of Exercise-Induced Muscle Damage Following Maximal Eccentric Contractions in Men and Boys. Pediatr Exerc Sci. 2017 Aug;29(3):316-325. doi: 10.1123/pes.2016-0185. Epub 2017 Feb 6. PMID 28165870
- [Background] Kyrolainen H, Avela J, McBride JM, Koskinen S, Andersen JL, Sipila S, Takala TE, Komi PV. Effects of power training on muscle structure and neuromuscular performance. Scand J Med Sci Sports. 2005 Feb;15(1):58-64. doi: 10.1111/j.1600-0838.2004.00390.x. PMID 15679573
- [Background] Ispirlidis I, Fatouros IG, Jamurtas AZ, Nikolaidis MG, Michailidis I, Douroudos I, Margonis K, Chatzinikolaou A, Kalistratos E, Katrabasas I, Alexiou V, Taxildaris K. Time-course of changes in inflammatory and performance responses following a soccer game. Clin J Sport Med. 2008 Sep;18(5):423-31. doi: 10.1097/JSM.0b013e3181818e0b. PMID 18806550
- [Background] Hughes JD, Massiah RG, Clarke RD. The Potentiating Effect of an Accentuated Eccentric Load on Countermovement Jump Performance. J Strength Cond Res. 2016 Dec;30(12):3450-3455. doi: 10.1519/JSC.0000000000001455. PMID 27100315
- [Background] Cormie P, McCaulley GO, Triplett NT, McBride JM. Optimal loading for maximal power output during lower-body resistance exercises. Med Sci Sports Exerc. 2007 Feb;39(2):340-9. doi: 10.1249/01.mss.0000246993.71599.bf. PMID 17277599
- [Background] Walker S, Blazevich AJ, Haff GG, Tufano JJ, Newton RU, Hakkinen K. Greater Strength Gains after Training with Accentuated Eccentric than Traditional Isoinertial Loads in Already Strength-Trained Men. Front Physiol. 2016 Apr 27;7:149. doi: 10.3389/fphys.2016.00149. eCollection 2016. PMID 27199764